CLINICAL TRIAL: NCT06712368
Title: Effect of Virtual Reality on Pain, Arterial Blood Gases and Functional Capacity in Children After Open Heart Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mamdouh Abdelmoaty Abdelaal, Demonstrator at Department of Pediatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005353
Record Dates: First submitted 2024-11-24; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Children After Open Heart Surgery
Keywords: virtual reality, heart surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Designed cardiac physical therapy program ( study group ) (Active Comparator): Designed cardiac physical therapy program
  Interventions: Other: Designed cardiac physical therapy program
- virtual reality group (study group) (Experimental): virtual reality glasses Designed cardiac physical therapy program applied through virtual reality glasses for study group
  Interventions: Device: virtual reality glasses

INTERVENTIONS:
Device: virtual reality glasses — Designed cardiac physical therapy program applied through virtual reality glasses for study group
  Other Names: Experimental: study group
  Arms: virtual reality group (study group)
Other: Designed cardiac physical therapy program — Designed cardiac physical therapy program without virtual reality glasses
  Arms: Designed cardiac physical therapy program ( study group )

SUMMARY:
This study will be conducted to investigate:

* The effect of virtual reality on pain in children after open heart surgery,
* The effect of virtual reality on arterial blood gases in children after open heart surgery,
* The effect of virtual reality on functional capacity in children after open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Both genders will be included.
* Their age range from 6 to 12 years.
* Children after open heart surgery ( phase I cardiac rehabilitation).

Exclusion Criteria:

The children have one or more of the following will be excluded:

* Any child Suffering from any other chronic congenital diseases.
* Severe visual or auditory problems.
* Neurological problems.
* Vertigo problems.
* Post surgical hemorrhage.
* Post surgical arrhythmia.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
pain | 1 hour /session 1 time / day for 5 consecutive days
  Pain assessment by Wong-Baker faces scale:
arterial blood gases | 1 hour /session 1 time / day for 5 consecutive days
  Arterial Blood Gases Analysis to detect blood gases
functional capacity | 1 hour /session 1 time / day for 5 consecutive days
  The Six-Minute Walk Test (6MWT) for assessment functional capacity

CONTACTS AND LOCATIONS:
Locations (1):
- National heart institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No